CLINICAL TRIAL: NCT01210105
Title: Comparison of Different Video Laryngoscopes in Ice-pick Position in an Manikin With Restricted Access to the Airway
Brief Title: Ice-pick Intubation With Video Laryngoscopes in a Manikin With Restricted Access to the Airway
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, J. Hinkelbein, PD Dr. med., University of Cologne
Other Study IDs: 10-182-3
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Tracheal Intubation
Keywords: intubation; video laryngoscopes

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Macintosh #3 Laryngoscope
- Glidescope
- Ambu Pentax AWS
- McGrath
- Airtraq
- Storz C-MAC

SUMMARY:
To determine whether video laryngioscopes facilitate intubation in ice-pick position in a manikin with restricted access to the airway

DETAILED DESCRIPTION:
To determine whether video laryngioscopes facilitate intubation in ice-pick position (also called inverse intubation) in a manikin with restricted access to the airway

ELIGIBILITY:
Inclusion Criteria:

* anaesthesiologists
* experienced in airway management
* experienced in emergency medicine

Exclusion Criteria:

* no experience in airway management
* missing infiormed consent

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: anaesthesiologists
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
tracheal intubation | max 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A Wetsch, MD, Principal Investigator — Department of Anaesthesiology, University of Cologne
Locations (1):
- Department of Anaesthesiology and Postoperative Critical Care, Cologne, Germany

REFERENCES:
- [Derived] Wetsch WA, Hellmich M, Spelten O, Schier R, Bottiger BW, Hinkelbein J. Tracheal intubation in the ice-pick position with video laryngoscopes: a randomised controlled trial in a manikin. Eur J Anaesthesiol. 2013 Sep;30(9):537-43. doi: 10.1097/EJA.0b013e3283614119. PMID 23736089